CLINICAL TRIAL: NCT02177305
Title: A Single Increasing Dose Tolerance Study After Ocular Administration of Tiotropium (Single Doses: 0.02 - 0.4 mcg) in Healthy Male Volunteers (Randomised, Placebo-controlled, Double-blind, Parallel Groups).
Brief Title: Dose Tolerance Study After Ocular Administration of Tiotropium in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.138
Record Dates: First submitted 2014-06-20; First posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Tiotropium dose group 1 (Experimental): 0.02 mcg tiotropium solution
  Interventions: Drug: 0.02 mcg tiotropium solution; Drug: Placebo solution
- Tiotropium dose group 2 (Experimental): 0.04 mcg tiotropium solution
  Interventions: Drug: 0.04 mcg tiotropium solution; Drug: Placebo solution
- Tiotropium dose group 3 (Experimental): 0.08 mcg tiotropium solution
  Interventions: Drug: 0.08 mcg tiotropium solution; Drug: Placebo solution
- Tiotropium dose group 4 (Experimental): 0.16 mcg tiotropium solution
  Interventions: Drug: 0.16 mcg tiotropium solution; Drug: Placebo solution
- Tiotropium dose group 5 (Experimental): 0.28 mcg tiotropium solution
  Interventions: Drug: 0.28 mcg tiotropium solution; Drug: Placebo solution
- Tiotropium dose group 6 (Experimental): 0.40 mcg tiotropium solution
  Interventions: Drug: 0.40 mcg tiotropium solution; Drug: Placebo solution

INTERVENTIONS:
Drug: 0.02 mcg tiotropium solution
  Arms: Tiotropium dose group 1
Drug: 0.04 mcg tiotropium solution
  Arms: Tiotropium dose group 2
Drug: 0.08 mcg tiotropium solution
  Arms: Tiotropium dose group 3
Drug: 0.16 mcg tiotropium solution
  Arms: Tiotropium dose group 4
Drug: 0.28 mcg tiotropium solution
  Arms: Tiotropium dose group 5
Drug: 0.40 mcg tiotropium solution
  Arms: Tiotropium dose group 6
Drug: Placebo solution

SUMMARY:
Safety and tolerability after ocular administration

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Age range from 21 to 50 years
* Within ± 20% of normal weight (Broca-Index)
* Written informed consent given

Exclusion Criteria:

* Results of the medical examinations or laboratory tests are judged by the clinical investigator to differ significantly from normal clinical values
* Volunteers with known gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Volunteers with disease of the central nervous system (such as epilepsy) or with psychiatric disorders
* Volunteers with known history of orthostatic hypotension, fainting spells or blackouts
* Volunteers with chronic or relevant acute infections
* Volunteers with history of allergy/ hypersensitivity (including drug allergy)
* Volunteers with known eye diseases (incl. glaucoma), with hyperopia (> 3 diopters) or with contact lenses
* Volunteers with intraocular pressure > 22 mmHg
* Volunteers with predisposition to narrow-angle glaucoma
* Volunteers with disturbed micturition
* Volunteers who have taken a drug with a long half-life (≥ 24 hours) within ten half-lives of the respective drug before enrolment in the study
* Volunteers who received any other drugs which might influence the results of the trial during the week previous the start of the study
* Volunteers who have participated in another study with an investigational drug within the last two months preceding this study
* Volunteers who smoke (> 10 cigarettes or 3 cigars or 3 pipes/day)
* Volunteers who are not able to refrain from smoking on study day
* Volunteers who drink more than 40 g of alcohol per day
* Volunteers who are dependent on drugs
* Volunteers who have donated blood (≥ 100 ml) within the last four weeks
* Volunteers who participated in excessive physical activities (e.g. competitive sports) within the last week before the study

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 1998-10; Primary Completion 1998-12 (Actual)

PRIMARY OUTCOMES:
Change in pupil diameter | baseline, after 24 hours
Change in pupillary reflex | baseline, after 24 hours
Change in intraocular pressure | baseline, after 24 hours
Change in accommodation | baseline, after 24 hours

SECONDARY OUTCOMES:
Change from baseline in blood pressure | on Day 1 before and 24 hours after treatment and within 8 days after treatment day
Change from baseline in pulse rate | on Day 1 before and 24 hours after treatment and within 8 days after treatment day
Change in 12-lead ECG | on Day 1 before and 24 hours after treatment and within 8 days after treatment day
Changes from baseline in standard laboratory examinations | Baseline and within 8 days after treatment day
Occurrence of Adverse Events | until 8 days after treatment day